CLINICAL TRIAL: NCT03148704
Title: Intensive Medicines Monitoring Project of Palonosetron Hydrochloride Capsules
Brief Title: Intensive Medicines Monitoring Project of Palonosetron Hydrochloride Capsules (Ruo Shan®)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Other Study IDs: Ruo Shan new drug monitoring
Record Dates: First submitted 2017-05-04; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Palonosetron
MeSH Terms: interventions — Palonosetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- palonosetron palonosetron hydrochloride: A continuous sequence of patients using palonosetron palonosetron hydrochloride capsules(Ruo Shan®)
  Interventions: Drug: palonosetron hydrochloride capsules

INTERVENTIONS:
Drug: palonosetron hydrochloride capsules — Collect all the patients' safty and efficacy data as long as they use palonosetron hydrochloride capsules(Ruo Shan®) .Specific methods of using the drugs are not limited .
  Other Names: Ruo Shan®

SUMMARY:
Observe palonosetron hydrochloride capsules'(Ruo Shan®) safety and efficacy information in the real world using.

DETAILED DESCRIPTION:
Observe palonosetron hydrochloride capsules'(Ruo Shan®) safety and efficacy information in the real world using.

1. Observe the adverse effects of palonosetron hydrochloride capsules(Ruo Shan®) that we already known, and whether there is any new adverse effects.Observe the incidence and the situation of adverse effects. Pay attention to the adverse effects in special groups, like pregnant women, children, elderly patients, and patients with liver and kidney dysfunction. Observe other safety issues related to drug using method, drug packaging method and drug quality.

   [Time Frame: A period between the first day of using Palonosetron Hydrochloride Capsules (Ruo Shan®) to the fifth day]

   Secondary Outcome Measures:
2. Furtherly clarify the efficacy of palonosetron hydrochloride capsules, and the widely used population characteristics, and clinical using features of palonosetron hydrochloride capsules.

[Time Frame: A period between the first day of using Palonosetron Hydrochloride Capsules (Ruo Shan®) to the fifth day]

ELIGIBILITY:
Inclusion Criteria:

* Use palonosetron hydrochloride capsules(Ruo Shan®) .Specific methods of using the drugs are not limited .
* Elderly patients do not need to adjust the dosage of the drug.
* Children using the drug and dose adjustment need to be evaluated by the doctor.
* Pregnant and lactating patients using the drug need to be evaluated by the doctor.
* 5-HT3RA allergic patients do not recommend the use of this drug.

Exclusion Criteria:

* All situations that the doctor think it is not suitable to use palonosetron hydrochloride capsules(Ruo Shan®) .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A continuous sequence of patients using palonosetron palonosetron hydrochloride capsules(Ruo Shan®)
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-03-08 (Estimated); Study Completion 2018-06-08 (Estimated)

PRIMARY OUTCOMES:
Report the palonosetron hydrochloride capsules'(Ruo Shan®) safety information in the real world using. | A period between the first day of using Palonosetron Hydrochloride Capsules (Ruo Shan®) to the fifth day
  1. Report the adverse effects of palonosetron hydrochloride capsules(Ruo Shan®) that we already known；
  2. Report if there is any new adverse effects；
  3. Report the incidence and the situation of the above adverse effects；
  4. Report the adverse effects in special groups, like pregnant women, children, elderly patients, and patients with liver and kidney dysfunction；
  5. Report other safety issues related to drug using method, drug packaging method and drug quality.

SECONDARY OUTCOMES:
Report the efficacy of palonosetron hydrochloride capsules. | A period between the first day of using Palonosetron Hydrochloride Capsules (Ruo Shan®) to the fifth day
  Report the control condition of nausea and vomiting.
Report the widely used population characteristics. | A period between the first day of using Palonosetron Hydrochloride Capsules (Ruo Shan®) to the fifth day
  Report the patients' disease, age, treatment, and chemotherapy drugs.
Report the clinical using features of palonosetron hydrochloride capsules. | A period between the first day of using Palonosetron Hydrochloride Capsules (Ruo Shan®) to the fifth day
  Report the Using does,time,and frequency of palonosetron hydrochloride capsules,and the concomitant drugs .

CONTACTS AND LOCATIONS:
Overall Officials: qin shu kui, Study Chair — The 81st Hostital of PLA
Locations (1):
- The 81st Hostital of PLA, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No